CLINICAL TRIAL: NCT00975806
Title: A Phase 1/2, Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Safety and Efficacy of Lenalidomide in Combination With Sunitinib in Subjects With Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Study of Lenalidomide in Combination With Sunitinib to Evaluate the Safety and Efficacy in Patients With Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: MTD determined sub-optimal as efficacious treatment for renal cell carcinoma.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-RCC-001
Record Dates: First submitted 2009-09-09; First posted 2009-09-11 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Lenalidomide; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Participants received an oral dose of lenalidomide MTD (mg) capsule administered in combination with a single dose of sunitinib 37.5 mg on days 1-21 of each 21-day cycle
  Interventions: Drug: Lenalidomide; Drug: Sunitinib
- Cohorts F and G (Experimental): Participants received an oral daily dose of lenalidomide on Days 1 to 21 in combination with a single oral daily dose of sunitinib 37.5 mg on days 1 to 14 or days 1 to 21 of each 21-day cycle
  Interventions: Drug: Lenalidomide; Drug: Sunitinib

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide MTD mg by mouth (PO) daily for Days 1- 21 in combination
  Other Names: CC-5013; Revlimid
Drug: Sunitinib — Sunitinib 37.5 mg PO daily on days 1-21 of each 21-day cycle in Cohort A or on days 1-14 in Cohorts F and G
  Other Names: Sutent

SUMMARY:
The purpose of this study was to determine the maximum tolerated dose, safety, and effectiveness of lenalidomide (CC-5013) administered in combination with sunitinib as treatment for patients with renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic Renal Cell Carcinoma.
2. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.

Exclusion Criteria:

1. Prior chemotherapy.
2. Prior treatment with lenalidomide, thalidomide, pomalidomide, or sunitinib.
3. Laboratory values outside normal ranges.
4. Myocardial infarction (MI) within past 12 months.
5. Current congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debora Barton, MD, Study Director — Celgene Corporation
Locations (3):
- United States (3):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Result] Rini B, Redman B, Garcia JA, Burris HA 3rd, Li S, Fandi A, Beck R, Jungnelius U, Infante JR. A phase I/II study of lenalidomide in combination with sunitinib in patients with advanced or metastatic renal cell carcinoma. Ann Oncol. 2014 Sep;25(9):1794-1799. doi: 10.1093/annonc/mdu212. Epub 2014 Jun 8. PMID 24914044

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg: Lenalidomide 10 mg and sunitinib 37.5 mg by mouth (PO) every day (QD) on Days 1 to 21 of each 21-day cycle
- Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg: Lenalidomide 10 mg PO QD on Days 1 to 21 and sunitinib 37.5 mg PO QD on Days 1 to 14 of each 21-day cycle
- Cohort G: Lenalidomide 15mg and Sunitinib 37.5mg: Lenalidomide 15 mg PO QD on Days 1 to 21 and sunitinib 37.5 mg PO QD on Days 1 to 14 of each 21-day cycle
Period: Overall Study
Arm/Group | Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg | Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg | Cohort G: Lenalidomide 15mg and Sunitinib 37.5mg
Started | 5 | 7 | 4
Completed | 0 (Participants were prematurely discontinued) | 0 (Participants were prematurely discontinued) | 0 (Participants were prematurely discontinued)
Not Completed | 5 | 7 | 4
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Disease Progression | 1 | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Physician decision and disease related | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population includes all participants who received at least one dose of study drug.
Groups:
- Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg: Lenalidomide 10 mg and sunitinib 37.5 mg PO QD on Days 1 to 21 of each 21-day cycle
- Total: Total of all reporting groups
Arm/Group | Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg | Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg | Cohort G: Lenalidomide 15mg and Sunitinib 37.5mg | Total
Number analyzed (Participants) | 5 | 7 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (18.84) | 57.1 (4.88) | 57.3 (5.62) | 56.5 (10.56)
Age, Customized [Number; unit: participants]
  ≤65 years | 4 | 7 | 4 | 15
  >65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 8
  Male | 3 | 3 | 2 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White) | 4 | 6 | 4 | 14
  Black or African American | 1 | 0 | 0 | 1
  Unknown | 0 | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis.
  0 = Fully Active (Most Favorable Activity)
  1. = Restricted activity but ambulatory
  2. = Ambulatory but unable to carry out work activities
  3. = Limited Self-Care
  4. = Completely Disabled, No self-care (Least Favorable Activity)
  participants
    0 = fully active | 4 | 4 | 4 | 12
    1 = restricted activity but ambulatory | 1 | 3 | 0 | 4
    3 (Limited Self-Care) | 0 | 0 | 0 | 0
    4 (Completely Disabled) | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD)
Description: The MTD of lenalidomide in combination with sunitinib was defined as the highest dose level at which no more than 1 out of 6 participants experienced a dose limiting toxicity (DLT). Dose limiting toxicities were:
  • Inability to deliver Lenalidomide in Cycle 1 due to a drug-related toxicity resulting in:
  * Grade (GR) 3 or 4 non-hematological toxicity lasting for ≥ 14 days
  * Febrile neutropenia
  * Gr 4 neutropenia lasting for ≥ 7 days
  * Gr 4 thrombocytopenia The occurrence of one of the above drug-related toxicities resulting in a clinical and/or laboratory assessment being done within 7 days following the initial finding to examine the participants for resolution of the toxicity. Lack of resolution of the toxicities was considered a DLT.
  If ≤ 7 doses of lenalidomide or Sunitinib were missed in Cycle 1 due to non-drug related event, the participant data was to be included in the evaluation of dose escalation.
Time Frame: Within 21 days of first dose of treatment
Population: Safety population includes all participants who received at least one dose of the study drug.
Measure: Number; unit: mg
Arm/Group | Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg
Number analyzed (Participants) | 16
mg | 10

2. Primary Outcome: Phase 2: Tumor Response Rate According to Response Evaluation Criteria In Solid Tumors (RECIST 1.1)
Description: Tumor response was to be evaluated every 3 cycles beginning with Cycle 3 Day 1 and at treatment discontinuation. Response was to be defined by RECIST 1.1 criteria:
  * Complete response-disappearance of all lesions
  * Partial response-30% decrease in the sum of diameters of target lesions from baseline
  * Stable disease-neither shrinkage nor increase of lesions.
  * Progressive Disease-20% increase in the sum of diameters of target lesions from nadir.
Time Frame: After at least 3 cycles of treatment
Population: Analysis was not performed due to the early termination of the study. The cumulative frequency and severity of toxicities observed at each dose level, including Maximum Tolerated Dose (MTD), were higher than expected and evident during all cycles and all dose levels in Phase 1. The decision was made not to open the Phase 2 portion of the study.
Groups:
- Phase 2: Lenalidomide 10mg and Sunitinib 37.5 mg: Lenalidomide 10 mg and sunitinib 37.5 mg by mouth (PO) every day (QD) on Days 1 to 21 of each 21-day cycle
Arm/Group | Phase 2: Lenalidomide 10mg and Sunitinib 37.5 mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) While on Both Lenalidomide and Sunitinib
Description: Adverse event (AE) = any noxious, unintended, or untoward medical occurrence occurring at any dose that may appear or worsen in a participant during the course of a study, including new intercurrent illness, worsening concomitant illness, injury, or any concomitant impairment of participants health, including laboratory test values, regardless of etiology. Serious adverse event (SAE) = any AE which: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. TEAE = any AE occurring or worsening on or after the first treatment with any study drug. Related = suspected by investigator to be related to study treatment. National Cancer Institute [NCI] Common Toxicity Criteria for Adverse Events [CTCAE], Version 4.0, grades: 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, 5 = death
Time Frame: First day of study drug to within 28 days after the last dose of the last study drug; The duration of exposure to lenalidomide and sunitinib was 7.0 to 327 and 7.0 to 328 days respectively
Population: Safety population includes all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg | Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg | Cohort G: Lenalidomide 15mg and Sunitinib 37.5mg
Number analyzed (Participants) | 5 | 7 | 4
participants
  Participants with at least 1 TEAE | 5 | 7 | 4
  Participants with at least 1 serious TEAE | 3 | 4 | 2
  ≥ 1 TEAE leading to stopping lenalidomide | 2 | 2 | 2
  ≥ 1 TEAE leading to stopping sunitinib | 2 | 2 | 2
  ≥ 1 TEAE -> dose reduction/interrruption of Len | 5 | 6 | 4
  ≥ 1 TEAE dose reduction/interrruption of Sunitinib | 5 | 5 | 3
  Participants with ≥1 TEAE related to lenalidomide | 5 | 7 | 4
  Participants with ≥1 TEAE related to Sunitinib | 5 | 7 | 4
  ≥ 1 NCI CTC Gr 3 or higher TEAE | 5 | 6 | 4
  ≥ 1 NCI CTC Gr 3 or higher related to lenalidomide | 4 | 5 | 4
  ≥ 1 NCI CTC Gr 3 or higher related to Sunitinib | 4 | 5 | 4
  ≥ 1 serious TEAE related to lenalidomide | 2 | 2 | 0
  ≥ 1 serious TEAE related to sunitinib | 1 | 2 | 2

4. Secondary Outcome: Phase 1 : Tumor Response Rate According to RECIST 1.1
Description: Tumor response was evaluated every 3 cycles beginning with Cycle 3 Day 1 and at treatment discontinuation. Response was evaluated using the Response Criteria Evaluation in Solid Tumors (RECIST 1.1) criteria:
  Treatment response includes both complete response and partial response
  * Complete response-disappearance of all lesions
  * Partial response-30% decrease in the sum of diameters of target lesions from baseline
  * Stable disease-neither shrinkage nor increase of lesions
  * Progressive Disease-20% increase in the sum of diameters of target lesions from nadir
Time Frame: Every 3 cycles; up to month 25
Population: Intent to Treat Population includes participants who took at least one dose of study drug. Study participants with stable disease also reported.
Measure: Number; unit: participants
Arm/Group | Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg | Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg | Cohort G: Lenalidomide 15mg and Sunitinib 37.5mg
Number analyzed (Participants) | 5 | 7 | 4
participants
  Complete Response | 0 | 0 | 0
  Partial Response | 1 | 0 | 0
  Stable Disease | 1 | 3 | 3

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival was defined as the time from the start of study drug therapy to the first observation of disease progression or death due to any cause, whichever came first.
Time Frame: Day 1 of study drug to disease progression or death
Population: Analysis was not performed due to the early termination of the study. The cumulative frequency and severity of toxicities observed at each dose level, including MTD, were higher than expected and evident during all cycles and all dose levels in Phase 1. The decision was made not to open the Phase 2 portion of the study.
Arm/Group | Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg | Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg | Cohort G: Lenalidomide 15mg and Sunitinib 37.5mg
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the initial response date to progressive disease (PD) for participants who achieved an objective confirmed complete response (CR) or partial response (PR)
Time Frame: Day 1 of initial response date to progressive disease
Population: as for outcome 2
Arm/Group | Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg | Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg | Cohort G: Lenalidomide 15mg and Sunitinib 37.5mg
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the start of study drug therapy to death.
Time Frame: Day 1 of study drug to death
Population: as for outcome 2
Arm/Group | Cohort A: Lenalidomide 10mg and Sunitinib 37.5 mg | Cohort F: Lenalidomide 10mg and Sunitinib 37.5mg | Cohort G: Lenalidomide 15mg and Sunitinib 37.5mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Phase 1 Only. From the date of the first study drug dose to within 28 days after the study drug treatment was discontinued.
Description: Median treatment duration with Lenalidomide and Sunitinib was shortest in Cohort A at 41 days (range = 17 to 189 days) and longest in Cohort G = 97 days (range: 60 to 125 days) of lenalidomide treatment and 97.5 days (range = 54 to 125 days) of Sunitinib
Groups:
- Cohort A: Lenalidomide 10 mg QD and sunitinib 37.5 mg QD on Days 1-21 of each 21-day cycle
- Cohort F: Lenalidomide 10 mg QD on Days 1-21 of each 21-day cycle and sunitinib 37.5 mg QD on Days 1-14 of each 21-day cycle
- Cohort G: Lenalidomide 15 mg QD on Days 1-21 of each 21-day cycle and sunitinib 37.5 mg QD on Days 1-14 of each 21-day cycle
Arm/Group | Cohort A | Cohort F | Cohort G
Serious Adverse Events (participants affected / at risk) | 3/5 | 4/7 | 2/4
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=5) | Cohort F (N=7) | Cohort G (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=5) | Cohort F (N=7) | Cohort G (N=4)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 2
Thrombocytpenia (Blood and lymphatic system disorders) | 2 | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Haemogloinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Splinter Haemorrhages (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0
Thyroiditis Subacute (Endocrine disorders) | 0 | 0 | 1
Lacrimation Increased (Eye disorders) | 1 | 1 | 0
Eye Swelling (Eye disorders) | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0
Tear discolouration (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 2
Nausea (Gastrointestinal disorders) | 4 | 4 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Tongue Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Tongue Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 7 | 4
Chills (General disorders) | 1 | 0 | 0
Mucosal Inflammation (General disorders) | 1 | 3 | 1
Non-cardiac Chest Pain (General disorders) | 1 | 1 | 1
Early Satiety (General disorders) | 0 | 1 | 0
Face Oedema (General disorders) | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 3 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1
Infected Bites (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 2 | 2 | 1
Transaminases Increased (Investigations) | 2 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 0 | 0
Neutrophil Count Decreased (Investigations) | 1 | 1 | 2
White Blood Cell Count Decreased (Investigations) | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 2
Blood Alkaline Phosphatase (Investigations) | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Decreasd Appetite (Metabolism and nutrition disorders) | 2 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 4 | 4 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 2
Headache (Nervous system disorders) | 2 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 1 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 1 | 1
Scrotal Oedema (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Orophryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Scar Pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Multicenter publications must include input from investigators and Celgene, and agreement be established before publication. Results from a center cannot be submitted for publication prior to a multicenter publication unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene ≤ 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to ≤ 90 days.